CLINICAL TRIAL: NCT03256591
Title: A Comparison of the Implementation of HBB Training Using Facilitators With and Without Simulation Methodology Training
Brief Title: Implementation of HBB Training With Facilitators That Have Undergone Simulation Methodology Training
Acronym: SimHBB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MUST 21/06-16c
Record Dates: First submitted 2017-08-15; First posted 2017-08-22 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Maternal Health; Newborn; Vitality

STUDY DESIGN:
Intervention Model Description: Investigators will conduct a prospective, randomized controlled trial to determine if the implementation of a simulation facilitator training program for HBB compared with no facilitator training in simulation is superior in terms of the acquisition of knowledge, acute care skills, and teamwork skills of pre-service medical students. Investigators will randomly randomly assign study participants to either intervention or control arm in a 1:1 ratio.
Masking Description: No masking will be done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBB plus simulation training (Experimental): Participants receive training from facilitators for HBB training with simulation skills
  Interventions: Other: HBB facilitators with simulation training
- Control (No Intervention): Participants receive training from facilitators for HBB training without simulation skills

INTERVENTIONS:
Other: HBB facilitators with simulation training — HBB training from facilitators with simulation skills. Standard HBB facilitators do not have simulation skills
  Arms: HBB plus simulation training

SUMMARY:
Helping Babies Breathe (HBB) implementation is associated with reduction in neonatal deaths and reduction in fresh stillbirths. HBB has successfully integrated some aspects of simulation into an educational curriculum that teach the management of neonatal emergencies in resource-constrained countries.

Simulation based training brings special advantages and may enhance HBB training. Critical elements of simulation such as enhanced realism and post-event debriefing may carry potential to strengthen HBB training to attain maximum impact. However, evidence for the effectiveness of this combined approach is limited.

DETAILED DESCRIPTION:
Helping Babies Breathe (HBB) implementation is associated with reduction in neonatal deaths and reduction in fresh stillbirths. HBB has successfully integrated some aspects of simulation into an educational curriculum that teach the management of neonatal emergencies in resource-constrained countries.

High levels of physical, emotional and conceptual realism are important features of simulation-based learning that impact learning outcomes. Formal debriefing is characterized as the most important element of simulation based education. Structured feedback in a safe learning environment provides the opportunity for learning of clinically relevant material. Guided reflection transfers the responsibility for learning to the participants and solidifies knowledge, skills and behaviors for transfer to clinical practice.

Simulation based training brings special advantages and may enhance HBB training. Critical elements of simulation such as enhanced realism and post-event debriefing may carry potential to strengthen HBB training to attain maximum impact. However, evidence for the effectiveness of this combined approach is limited.

ELIGIBILITY:
Inclusion Criteria:

* Only trained facilitators are eligible to participate
* Must hold a Faculty position or are a health care provider at KIU Teaching Hospital in western Uganda
* Are engaged in teaching health students.
* Participating medical students are those enrolled at KIU Teaching Hospital in western Uganda

Exclusion Criteria:

* Faculty and hospital workers who are not engaged in teaching health students.
* Medical students not enrolled at KIU Teaching Hospital, western Uganda

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge | Change in knowledge scores at 6 months from Baseline
  The primary outcome for this analysis is level of knowledge. For each course, learners will be assessed at baseline and at course-end to determine their knowledge via multiple choice test. Scores out of 100% will be computed

SECONDARY OUTCOMES:
Clinical skills | Change in clinical skills at 6 months from baseline
  The clinical skills outcome (via short neonatal resuscitation simulation scenario - HBB OSCE B). HBB OSCE B assessment will be conducted by the facilitator.
Facilitator debriefing skills | Change in facilitator skills at 6 months from baseline
  Facilitator debriefing skills will be assessed using the OSAD. OSAD assessments will be conducted by a pre-trained rater who will rate facilitator performance in real time.

CONTACTS AND LOCATIONS:
Overall Officials: Santorini Data, MD, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Kampala International University, Ishaka, Bushenyi, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after appropriate permissions have been obtained.